CLINICAL TRIAL: NCT04531943
Title: Feminizing Hormone Therapy and the Rectal Mucosa Immune Environment in Transgender Women
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Colleen Kelley, Associate Professor, Emory University
Other Study IDs: IRB00112414; R01AI147839 (NIH); R21AI157911 (NIH)
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-06

CONDITIONS: HIV Prevention
Keywords: Transgender women
MeSH Terms: interventions — Estrogens; Progesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood and rectal mucosa samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- TGWSM Using Estrogen: Cohort 1 participants are in the cross-sectional study and will attend two study visits, participating in study activities for up to 12 weeks. Blood samples and rectal mucosal samples will be obtained. This group of participants in Cohort 1 consists of TGWSM currently using feminizing hormone therapy consisting of only estrogen.
  Interventions: Drug: Estrogen
- TGWSM Using Estrogen plus Progesterone: Cohort 1 participants are in the cross-sectional study and will attend two study visits, participating in study activities for up to 12 weeks. Blood samples and rectal mucosal samples will be obtained. This group of participants in Cohort 1 consists of TGWSM currently using feminizing hormone therapy consisting of estrogen and progesterone.
  Interventions: Drug: Estrogen plus Progesterone
- Cisgender MSM: Cohort 1 participants are in the cross-sectional study and will attend two study visits, participating in study activities for up to 12 weeks. Blood samples and rectal mucosal samples will be obtained. This group of participants in Cohort 1 consists of cisgender MSM.
- TGWSM Initiating Feminizing Hormone Therapy: Cohort 2 participants are in the longitudinal portion of the study and are TGWSM who are planning to initiate feminizing hormone therapy. Individuals in Cohort 2 will participate in study activities for 18 months.
  Interventions: Drug: Estrogen; Drug: Estrogen plus Progesterone

INTERVENTIONS:
Drug: Estrogen — Feminizing hormone therapy consisting of estrogen alone, as prescribed by the participant's healthcare provider.
  Groups: TGWSM Initiating Feminizing Hormone Therapy; TGWSM Using Estrogen
Drug: Estrogen plus Progesterone — Feminizing hormone therapy consisting of estrogen and progesterone, as prescribed by the participant's healthcare provider.
  Groups: TGWSM Initiating Feminizing Hormone Therapy; TGWSM Using Estrogen plus Progesterone

SUMMARY:
The overarching goal of this research study is to achieve a better understanding of the rectal mucosal effects of feminizing hormones in people assigned male sex at birth and currently taking feminizing hormones who have sex with men. Better understanding the rectal mucosa in this population will allow for the optimization of current biomedical HIV prevention interventions and enhance design of future interventions, including an effective HIV vaccine. This study will recruit approximately 520 transgender women who have receptive anal intercourse with men (TGWSM) and cis-gender men into one of two cohorts. Cohort 1 is a cross-sectional study and Cohort 2 is a longitudinal study; enrollment into each cohort is based on participant characteristics.

DETAILED DESCRIPTION:
Transgender women who have receptive anal intercourse with men (TGWSM; assigned male sex at birth and taking/planning to take feminizing hormone therapy) are at high risk of HIV, and many HIV infections occur due to exposure to the rectal mucosa. In this study, the researchers will examine the biologic effects of feminizing hormone therapy on the mucosal immune milieu of the rectum. A better understanding of rectal HIV transmission among TGWSM will lead to the development of improved biomedical prevention interventions.

Historically, TGWSM have been grouped with men who have sex with men (MSM) in HIV prevention studies due to presumed similar risks of rectal HIV exposure despite their unique psychosocial, biologic, and prevention needs. From a biologic perspective, many TGWSM use feminizing hormone therapy with uncertain rectal mucosal effects. The effects of endogenous and exogenous hormones in the human and animal-model female genital tract has been described with estrogen generally being seen as hindering HIV transmission and progesterone facilitating transmission; however, few studies report effects on the rectal mucosa. In addition, the intestinal mucosa is known to be steroidogenic, and colonic epithelial cells express estrogen receptor β, suggesting that exogenous hormone therapy likely has an effect on the rectal mucosa that could influence HIV transmission. For this project, the researchers will build upon our successful translational mucosal immunology program with a highly successful clinical research and retention infrastructure that was designed to understand factors that may influence rectal HIV transmission and propose to examine the effects of feminizing hormone therapy on the rectal mucosal resident cellular populations, transcriptome, and microbiome in TGWSM. In the rectal mucosa, the researchers will compare HIV target cell availability, the transcriptome, and microbiome in a cross-sectional cohort of 1) TGWSM on using feminizing hormone therapy (n=300) and 2) cisgender MSM (n=150). The researchers will also examine HIV target cell availability, the transcriptome, and microbiome in a longitudinal study of TGWSM (n=70) before and after initiating feminizing hormone therapy.

Two cohorts of HIV-negative TGWSM will be enrolled in this study. Cohort 1 will be a cross-sectional study where the researchers will enroll 300 TGWSM who are on feminizing hormone therapy and a control group of 150 sexually active cisgender men (assigned male sex at birth and currently identify as male) who have sex with men. Individuals in Cohort 1 will participate in study activities for up to 12 weeks. Cohort 2 is a longitudinal study where 70 TGWSM who are naïve to feminizing hormone therapy or have not taken feminizing hormone therapy for > 6 months and plan to initiate feminizing hormone therapy will be enrolled. Individuals in Cohort 2 will participate in study activities for 18 months.

ELIGIBILITY:
INCLUSION CRITERIA

Cohort 1, TGWSM using feminizing hormone therapy

* Assigned male sex at birth and currently using feminizing hormone therapy
* Aged 18-59 years
* Able to provide informed consent in the official language of the study site's country
* HIV negative
* Taking feminizing hormone therapy for at least the last 6 months with no change in dose for the last 3 months (i.e. no increase or decrease)

  * Feminizing hormone therapy is defined as use of oral, patch, topical, or injection estrogen therapy with or without progesterone therapy in people who were assigned male sex at birth but take feminizing hormones to affirm their current gender identity

    * Approximately half of the cohort to be using estrogen therapy alone and half using estrogen+progesterone
  * Anti-androgen therapy is permissive, but dose must also be stable for the last 3 months at the time of enrollment
* Willing to undergo peripheral blood and rectal biopsy sampling
* Willing to abstain from receptive anal intercourse for 72 hours before and for 1 week after rectal biopsy procedure
* Willing to answer sexual behavior questions

Cohort 1, Cisgender Males

* Assigned male sex at birth, currently identify as male gender (i.e. cisgender), man who has sex with men aged 18-59 years
* Able to provide informed consent in the official language of the study site's country
* HIV negative
* Receptive anal intercourse with a person assigned male sex at birth at least once in lifetime
* No history of taking supplemental steroids including testosterone replacement therapy in the last 12 months
* Willing to undergo peripheral blood and rectal biopsy sampling
* Willing to abstain from receptive anal intercourse for 72 hours before and for 1 week after rectal biopsy procedure.
* Willing to answer sexual behavior questions.

Cohort 2, Longitudinal study with TGWSM planning to initiate feminizing hormone therapy

* Assigned male sex at birth with plans to start feminizing hormone therapy
* Aged 18-59 years
* Able to provide informed consent in the official language of the study site's country
* Naïve to feminizing hormone therapy or no use in the last 6 months, including anti-androgen therapy.
* HIV negative
* Plans to initiate feminizing hormone therapy in next 6 months.

  * Feminizing hormone therapy is defined as use of oral, patch, topical, or injection estrogen therapy with or without progesterone therapy in people who were assigned male sex at birth but take feminizing hormones to affirm their current gender identity.
  * Anti-androgen therapy is permissive, but participants must also be initiating estrogen therapy to be eligible.
* Willing to undergo peripheral blood and rectal biopsy sampling
* Willing to abstain from receptive anal intercourse for 72 hours before and for 1 week after rectal biopsy procedure.
* Willing to answer sexual behavior questions.

EXCLUSION CRITERIA

* History of inflammatory bowel disease or other inflammatory, infiltrative, infectious or vascular condition involving the lower gastrointestinal tract that, in the judgment of the investigators, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel
* Significant laboratory abnormalities at baseline visit for rectal biopsies, including but not limited to:

  * Hemoglobin (Hgb) ≤ 10 g/dL
  * Partial thromboplastin time (PTT) > 1.5x upper limit of normal (ULN) or international normalised ratio (INR) > 1.5x ULN
  * Platelet count <100,000
* Any known medical condition that, in the judgment of the investigators, increases the risk of local or systemic complications of endoscopic procedures or pelvic examination, including but not limited to:

  * Uncontrolled or severe cardiac arrhythmia
  * Recent major abdominal, cardiothoracic, or neurological surgery in the last 12 months
  * History of uncontrolled bleeding diathesis
  * History of colonic, rectal, or vaginal perforation, fistula, or malignancy
  * History or evidence on clinical examination of ulcerative, suppurative, or proliferative lesions of the anorectal mucosa.
* Use of systemic (oral/IV) antibiotics within the 4 weeks prior to rectal mucosal sampling.

  * Participants may be screened/enrolled who do not meet this criterion, but rectal mucosal sampling will be deferred for at least 4 weeks from last systemic antibiotic use.
* Continued need for, or use during the 14 days prior to enrollment, of the following medications:

  * Aspirin or more than 4 doses of nonsteroidal anti-inflammatory drugs (NSAIDs)
  * Warfarin, heparin (low-molecular weight or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
  * Any form of rectally administered agent besides products (lubricants or douching) used for sexual intercourse
* Continued need for, or use during the 90 days prior to enrollment, of the following medications:

  * Systemic immunomodulatory agents
  * Supraphysiologic doses of steroids with the exception of short course steroids <7 days duration at the discretion of the investigator and feminizing hormone therapy as detailed in inclusion criteria
  * Experimental medications, vaccines, or biologicals
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants are assigned male sex at birth and currently using feminizing hormones (Cohort 1, Group 1) or planning to begin using feminizing hormones (Cohort 2). Cisgender males are also enrolling.
Study Population: A total of 520 HIV-negative TGWSM and cisgender MSM will be enrolled into one of two cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Percent of Rectal Mucosal Cluster of Differentiation 4 (CD4+) T Cells Expressing C-C Chemokine Receptor Type 5 (CCR5) in Cohort 1 | Day 1 (day of rectal mucosal sampling)
  The median percentage of rectal mucosal CD4+ T cells that express CCR5 will be compared between groups in Cohort 1.
Change in Percent of Rectal Mucosal CD4+ T cells expressing CCR5 in Cohort 2 | Baseline and up to 12 months after initiation of feminizing hormone therapy
  The median percentage of rectal mucosal CD4+ T cells that express CCR5 will be compared in Cohort 2, before hormone therapy begins and after hormone therapy.
Production of p24 from Rectal Mucosal Explant Challenge in Cohort 1 | Day 1 (day of rectal mucosal sampling)
  The median production of p24 from rectal mucosal explant challenge experiments as measured by the area under the curve will be compared between groups in Cohort 1.
Change in Production of p24 from Rectal Mucosal Explant Challenge in Cohort 2 | Baseline and up to 12 months after initiation of feminizing hormone therapy
  The median production of p24 from rectal mucosal explant challenge experiments as measured by the area under the curve will be compared in Cohort 2, before hormone therapy begins and after hormone therapy.
Relative abundance of Prevotellaceae in Cohort 1 | Day 1 (day of rectal mucosal sampling)
  The median relative abundance of Prevotellaceae measured from rectal mucosal secretions will be compared between groups in Cohort 1.
Change in Relative abundance of Prevotellaceae in Cohort 2 | Baseline and up to 12 months after initiation of feminizing hormone therapy
  The median relative abundance of Prevotellaceae measured from rectal mucosal secretions will be compared in Cohort 2, before hormone therapy begins and after hormone therapy.
Relative abundance of Bacteroidaceae in Cohort 1 | Day 1 (day of rectal mucosal sampling)
  The median relative abundance of Bacteroidaceae measured from rectal mucosal secretions will be compared between groups in Cohort 1.
Change in Relative abundance of Bacteroidaceae in Cohort 2 | Baseline and up to 12 months after initiation of feminizing hormone therapy
  The median relative abundance of Bacteroidaceae measured from rectal mucosal secretions will be compared in Cohort 2, before hormone therapy begins and after hormone therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published for this study (including text, tables, figures, and appendices), will be made available for sharing, after de-identification.
Supporting Information: Study Protocol
Time Frame: Data will be made available to researchers providing a methodologically sound proposal, beginning 9 months and ending 36 months following publication.
Access Criteria: Proposals should be directed to colleen.kelley@emory.edu. To gain access, data requestors will need to sign a data access agreement.